CLINICAL TRIAL: NCT00655005
Title: Investigation of Pain and Symptom Burden in Patients With Newly Diagnosed Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine; Director, Cancer Supportive Care Program; Director, Head and Neck Research Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC SUPP 0723; VU-VICC-SUPP-0723; VU-VICC-070493
Record Dates: First submitted 2008-04-08; First posted 2008-04-09 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire administration — Newly diagnosed HNC patients
  Other Names: Non specified
Procedure: quality-of-life assessment — following treatment
  Other Names: Non specified

SUMMARY:
RATIONALE: Collecting information by questionnaire about the quality of life of patients with head and neck cancer may help doctors learn more about the disease.

PURPOSE: This clinical trial is testing a questionnaire for assessing pain control, head and neck symptoms, and general symptoms of illness, demographics, moods, alcohol and tobacco history, and quality of life related to cancer in patients with newly diagnosed head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To pilot test a questionnaire measuring the collection of the following data from patients with newly diagnosed head and neck cancer: head and neck cancer-related symptoms, general demographics, pain control, general symptoms, mood, smoking and drinking history, and quality of life.
* To identify questions that may be unclear or difficult for patients to understand.
* To determine the time required for each patient to complete the questionnaire and assess the feasibility and burden to the patient.
* To determine the baseline incidence of symptoms and psychosocial issues in these patients.

OUTLINE: Patients complete a timed questionnaire comprising questions of head and neck symptoms, demographic information, pain control, symptom control, mood, smoking and drinking history, and anxiety and depression under the supervision of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of head or neck carcinoma

  * Newly diagnosed disease
* Able to speak English
* Able to give informed consent

Exclusion Criteria:

Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed HNC patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Pilot questionnaire testing of related symptoms, general demographics, pain control, general symptoms, mood, smoking and drinking history, and quality of life | at time of patient exam
  collection of the following data from newly diagnosed HNC patients:
  * head and neck cancer-related symptoms • general demographics • pain control
  * general symptoms • mood • smoking and drinking history • quality of life
  Questions will be identified that may be unclear or difficult for patients to understand for future revision.

SECONDARY OUTCOMES:
Time required for questionnaire completion by each patient | at time of patient exam
  The investigator will verbally explain the purpose of the study using a script (provided with this packet) and obtain verbal consent from the patient. The questionnaire will be handed to the patient with instructions on how to complete it. The investigator will remain available in the room to address any concerns regarding the questionnaire and to time how long the patient takes to complete the survey.
  When the patient has completed the questionnaire, the investigator will review it for completeness with the patient. The patient's participation in the study ends at this time.
Feasibility and patient burden assessment | at time of patient exam
Baseline incidence of symptoms and psychosocial issues | at time of patient exam

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States